CLINICAL TRIAL: NCT03551301
Title: Transitional Case Management for Patients Suffering From Substance Use Disorders
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Louise Penzenstadler, Principal investigator, University Hospital, Geneva
Other Study IDs: ID 2017-00733
Record Dates: First submitted 2018-04-24; First posted 2018-06-11 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Substance Use Disorders
Keywords: Substance Use Disorders; Case Management; Community Treatment; Hospital discharge
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transitional Case Management — TCM program is a type of very flexible community treatment in terms of frequency and intensity of care. This is facilitated by a small case load ratio per health care professional (1:10). The healthcare workers are specialised in SUD treatment. The intervention begins during hospitalisation and lasts around 4 weeks after discharge from the hospital.
  The main aim of this intervention is to accompany the patient in the difficult phase of transition between hospital and outpatient care and ensure their adherence to the treatment program. The healthcare workers will explore specific patient needs and ensure that health and social services are better coordinated to fit their needs. Another important aim is to reduce the number of (unplanned) hospitalizations and emergency room visits.

SUMMARY:
According to the World Health Organization the population suffering from addiction problems is increasing. This population is characterized by multiple needs at the medico-psychosocial level. However, some of these patients, a particular subgroup that we are going to be interested in the so-called "high need" user group, find it difficult to access and stay in outpatient treatment programs. They often present a chaotic use of the health system, including a high number of hospitalizations in times of crisis. They also show very low utilization of health care services, accompanied by social marginalization. This can be related to relapses and poor social functioning. A high number of relapses occur particularly at the end of hospitalization. Interventions in the field of addiction, such as Transitional Case Management (TCM) should increase the adherence of these patients to treatment by accompanying them in the sensitive period following hospitalization. One of the objectives of the study is to evaluate the impact of TCM on the number, duration and type of hospitalizations, as well as the number of emergency room visits. The investigators will also measure the duration until the possible future hospitalization, after the TCM. The secondary objectives of this study will be to see the effect of TCM on adherence to outpatient treatment. The investigators will focus on the impact of follow-up on the participant's medico-psycho-social network, substance use and other psychological variables. The investigators will also evaluate his or her psychiatric symptoms and global and social functioning. Life satisfaction and satisfaction with the care received will also be measured. The investigators will compare the population treated by the TCM with the other users of the addiction service who are hospitalized. The study will investigate this through questionnaires at the beginning of care, at one month, three months, six months and 12 months after the start of TCM management.

ELIGIBILITY:
Inclusion Criteria:

* Substance use disorder
* Hospitalisation at recruitment
* Substance Use Disorder according to the DSM-5 and one of the following criteria:
* No preexisting outpatient follow-up care or regular follow-up care
* More than three emergency room visits during the last 12 months
* More than three hospitalizations in psychiatric hospital during the last 12 months
* More than 40 hospitalization's days during the last 12 months
* First hospitalization for a SUD

Exclusion Criteria:

* Evidence of organic brain disease or learning disability based on the chart review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subgroup of high need users hospitalized in our addiction unit
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Hospital days | at 12 months
  Number of days in hospital

SECONDARY OUTCOMES:
Service use | at 12 months
  Number of hospital admissions
Patient network | 0, 3, 6, 12 months
  Number of persons in network
Time to first readmission to hospital | 0, 1, 3, 6, 12 months
  Number of days to first readmission
Type of admission (planned versus unplanned) | 0, 1, 3, 6, 12 months
  Type of admission (planned versus unplanned) reviewed on patient file
Number of ER visits | 0, 1, 3, 6, 12 months
  Number of ER visits reviewed on patient file
Treatment adherence | 0, 1, 3, 6, 12 months
  percentage of attended outpatient appointments reviewed on patient file
Number or Transitional Case Management interventions | 0, 1, 3, 6, 12 months
  Number or Transitional Case Management interventions
Addictive behaviour | 0, 1, 3, 6, 12 months
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST. V.3 French)
General psychiatric symptoms | 0, 1, 3, 6, 12 months
  Health of Nation Outcome Scale - French version (HoNOS-F): scores 0 - 52 (higher score = more psychiatric symptoms)
Global functioning | 0, 1, 3, 6, 12 months
  World Health Organization Disability Assessment Schedule (WHODAS)
General life satisfaction | 0, 1, 3, 6, 12 months
  Satisfaction With Life Scale: scores 5 - 35 (higher score = higher life satisfaction)
Advance directives written by the participants | at Baseline
  Advance directives written by the participant (yes - no)

OTHER OUTCOMES:
Patient satisfaction with Transitional Case Management | at 1 month
  Patient satisfaction with Transitional Case Management
Duration and intensity of Transitional Case Management intervention | at 1 month
  Daily contact log (Relevé quotidien des contacts (RQC))

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'addictologie HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chatton A, Khazaal Y, Penzenstadler L. A 13-item Health of the Nation Outcome Scale (HoNOS-13): validation by item response theory (IRT) in patients with substance use disorder. Addict Sci Clin Pract. 2023 Oct 24;18(1):64. doi: 10.1186/s13722-023-00416-8. PMID 37876018